CLINICAL TRIAL: NCT02472847
Title: Cannabinoid Control of Fear Extinction Neural Circuits in Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, K. Luan Phan, MD, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012-0242; R21MH093917 (NIH)
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Participants
Keywords: Marinol; Dronabinol; Fear extinction; Healthy volunteers
MeSH Terms: interventions — Dronabinol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): In a randomized, double-blind, placebo-controlled, between-subjects design, the investigators will couple a standard Pavlovian fear extinction paradigm in fMRI with an acute pharmacological challenge with oral dronabinol (synthetic THC) or placebo 2 hours prior to extinction learning in healthy adult volunteers and test extinction retention and maintenance 24 hours and 1 week later, respectively, after extinction learning.
  Interventions: Drug: Placebo
- Dronabinol (Active Comparator): In a randomized, double-blind, placebo-controlled, between-subjects design, the investigators will couple a standard Pavlovian fear extinction paradigm in fMRI with an acute pharmacological challenge with oral dronabinol (synthetic THC) or placebo 2 hours prior to extinction learning in healthy adult volunteers and test extinction retention and maintenance 24 hours and 1 week later, respectively, after extinction learning
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — Dronabinol (7.5mg) is administered only once by the oral route and is placed in opaque capsules with dextrose filler. Half of the participants will receive dronabinol.
  Other Names: Marinol
  Arms: Dronabinol
Drug: Placebo — Placebo is administered only once by the oral route and contains only dextrose in opaque capsules. Half of the participants will receive placebo.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The goal of the current proposal is to investigate the effects of a cannabinoid drug on the memory of extinguished fear in humans and the brain circuitry important for the recall of extinction learning. The investigators findings will translate previous discoveries from animal studies to humans and increase their understanding of the neurobiological mechanisms supporting retention of extinction memory. This proof-of-concept study is a critical translational first step towards the development of cannabinoid modulators as an adjunctive strategy to exposure-based therapies to augment extinction learning and prevent the return of fear memories in patients with post-traumatic stress and other anxiety disorders.

DETAILED DESCRIPTION:
The inability to suppress inappropriate fear responses is the hallmark of anxiety disorders, such as posttraumatic stress disorder (PTSD), panic, and phobia disorders. Extinction of fear occurs during exposure therapy; however, this is temporary and fear often re-emerges with the passage of time (spontaneous recovery), undermining the maintenance of therapeutic gains. Enhancing the neural and neurochemical substrates involved in retention of extinction memory will be critical to solving this challenge. Animal studies have shown that activation of the cannabinoid system within the amgydala, hippocampus, and ventromedial prefrontal cortex (AMYG, HPC, vmPFC, respectively), brain structures critical to fear expression and extinction learning, enhances fear extinction and its retention. Specifically, CB1 receptor agonists, such as Δ9-tetrahydrocannibinol (THC), can facilitate extinction recall by preventing recovery of extinguished fear in rats. However, this phenomenon has not been, but should be, investigated in humans. This proof-of-concept project specifically aims to assess the effects of THC on the recall of extinction learning and underlying neural circuit activation (HPC, vmPFC) when tested 24 hours and 1 week after extinction training, and to determine if the maintenance of extinction retention (1 week later) is mediated by the enhancement of vmPFC-HPC activation by THC observed during a recall test 24 hours after extinction learning. In a randomized, double-blind, placebo-controlled, between-subjects design, the investigators will couple a standard Pavlovian fear extinction paradigm in fMRI and simultaneous skin conductance recordings with an acute pharmacological challenge with oral, synthetic THC prior to extinction learning in healthy adult volunteers (n=80) and test extinction retention and maintenance of extinction learning at 24 hours and 1 week later, as well as fear renewal. This proof-of-concept study provides the most translational, impactful, informative, and critical test and first step towards the development of cannabinoid modulators as an adjunctive strategy to exposure-based therapies to augment extinction retention and prevent the return of fear memories in patients with PTSD and other anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

1. age 21-45
2. right-handed
3. free of lifetime diagnosis of Axis I psychiatric disorder
4. must be able to given informed consent
5. must be medically and neurologically healthy.

Exclusion Criteria:

1. any current medical condition requiring psychoactive/psychotropic medication or medication that would interact with dronabinol or interfere with study procedures
2. current or past allergic or adverse reaction or known sensitivity to cannabinoid-like substance (Dronabinol /Marijuana/Cannabis/THC, cannabinoid oil, sesame oil, gelatin, glycerin, and titanium dioxide.)
3. any current or past Axis I psychiatric disorder, including alcohol/substance abuse or dependence disorder
4. less than a high school education
5. lack of fluency in English
6. night shift work
7. currently pregnant or planning pregnancy or lactating (women)
8. unwilling/unable to sign informed consent document
9. inability to tolerate small, enclosed spaces without anxiety (e.g. claustrophobia), as determined by self-report and a preliminary session in a mock scanner
10. left-handed
11. presence of ferrous-containing metals within the body (e.g., aneurysm clips,shrapnel/retained particles)
12. under 21 or over 45 years of age
13. anticipation of a required drug test in the 4 weeks following the study. No vulnerable participant populations will be included in this study
14. participation in an experiment involving shocks in the last 6 months.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed initial screening visit, signed consent, if eligible scheduled for 4 fMRI scans. Participants were randomized immediately before the 2nd fMRI scan. Reasons for exclusion prior to randomization: 6 excluded during initial screening, 13 lost to follow up, 5 did not want to take study drug, 11 had scheduling conflicts.
Period: Overall Study
Arm/Group | Placebo | Dronabinol
Started | 24 | 26
Completed | 23 | 21
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dronabinol | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Customized [Number; unit: participants] — Between 21-45 years
  participants
    21-45 Years | 24 | 26 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 10 | 12
  Not Hispanic or Latino | 22 | 16 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 2 | 4
  White | 11 | 9 | 20
  More than one race | 1 | 7 | 8
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: BOLD Signal Measured by Functional Magnetic Resonance Imaging (fMRI)
Description: Mean BOLD hippocampal signal during extinction learning and retention task in brain responsebetween the placebo (PBO) and the dronabinol (THC) group. Target areas are analyzed from fMRI scans. The scans were completed on days 1, 2, 3, and 9. Participants were randomized to the PBO and THC condition and received either placebo or dronabinol on day 2, 2 hours prior to extinction learning. Data from days 1, 2, 3, & 9 was combined and a single value was averaged for each group.
Time Frame: Day 1, 2, 3, & 9
Population: The number of participants analyzed is 22 in the placebo group and 18 in the dronabinol group. The total number of participants who completed all 4 scanning sessions is 44. 4 participants were excluded from data analysis due to having poor quality fMRI data from any of the four sessions.
Measure: Mean (Standard Deviation); unit: parameter estimates (arbitrary units)
Arm/Group | Placebo | Dronabinol
Number analyzed (Participants) | 22 | 18
parameter estimates (arbitrary units) | 0.1631 (0.16784) | 0.5079 (0.30082)

ADVERSE EVENTS:
Arm/Group | Placebo | Dronabinol
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No